CLINICAL TRIAL: NCT03607149
Title: Pemetrexed in Maintenance in Patients With Impaired Renal Function: Randomized Phase 4 Multicenter Study Comparing 2 Dose Calculation Strategies (PKAPIR)
Brief Title: Pemetrexed in Maintenance in Patients With Impaired Renal Function, 2 Dose Calculation Strategies
Acronym: PKAPIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-002552-24
Record Dates: First submitted 2017-06-21; First posted 2018-07-31 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Pemetrexed; Non-small cell lung cancer; Clearance of creatine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STANDARD ARM (Active Comparator): Calculation of the dose of pemetrexed as a function of body surface area
  Interventions: Drug: Pemetrexed
- EXPERIMENTAL ARM (Experimental): Calculation of the pemetrexed dose as a function of the Clearance of creatine (CrCLCG)
  Interventions: Drug: Pemetrexed

INTERVENTIONS:
Drug: Pemetrexed — standard arm : calculating the dose of pemetrexed according to body surface area
  experimental arm: calculation of the dose of pemetrexed as a function of creatinine clearance (CrCLCG)

SUMMARY:
Pemetrexed is used in the treatment of non-small cell lung cancer (NSCLC). Its elimination is mainly renal and its nephrotoxicity requires an interruption of treatment when the CrCLCG falls below 45 mL / min. Patients with NSCLC frequently have impaired renal function by other cytotoxic drugs.

The dose adjustment of pemetrexed is performed as a function of body surface area (SC) without any pharmacokinetic rational. The challenge is to treat patients with renal insufficiency (RR) with a safe dose, based on CRCL, providing equivalent biological exposure to patients with preserved renal function.

DETAILED DESCRIPTION:
* Primary objective: Evaluate the impact of calculating the dose of pemetrexed to be administered versus creatine clearance according to Cockcroft-Gault (CrCLCG) versus body surface area (SC) on median time before discontinuation of treatment for renal function ≤ 45mL / min in patients treated for non-small cell lung cancer predominantly non-squamous in maintenance.
* Secondary objective: To evaluate the impact of calculating the dose of pemetrexed to be administered versus CRCLCG versus SC over time to treatment discontinuation, progression-free survival (PFS), and patient overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age
* Patient with non-small cell lung cancer predominantly non-epidermoid histologically documented
* Patient who is scheduled to initiate treatment or undergoing maintenance therapy by pemetrexed
* Neutrophils> 1500 / mm3; Chips> 100,000 / mm3
* Informed, dated and signed consent For patients of childbearing age, effective contraceptive method
* Creatinine clearance according to the Cockcroft-Gault formula between 70 and 45 mL / min
* PS = 0 or 1

Exclusion Criteria:

* Patient with a contraindication to pemetrexed therapy
* Patient with symptomatic brain metastases
* Pregnant or nursing women
* Patient under guardianship or curatorship or subject to a system of protection for persons of full age
* Patient not affiliated to a social security scheme (beneficiary or beneficiary)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2020-02-20 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Median time until treatment is stopped due to renal function ≤ 45mL / min | 1 year
  From date of randomization until the date of treatment is stopped

SECONDARY OUTCOMES:
Progression-free survival | up to 100 weeks
  From date of randomization until the date of death from any cause

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - CH William Morey, Chalon-sur-Saône
  - Centre Georges Francois Leclerc, Dijon
  - Centre Universitaire Hospitalier de Dijon, Dijon